CLINICAL TRIAL: NCT03235258
Title: ANRS CO10 EPF - Cohort of HIV-infected Children
Brief Title: Cohort of HIV-infected Children
Acronym: EPF
Status: Completed | Type: Observational
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: ANRS CO10 EPF
Record Dates: First submitted 2016-09-29; First posted 2017-08-01 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Children Infected by HIV
Keywords: HIV Infection; Adolescent
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 1 to 3 mL whole blood - 1 to 3mL plasma
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to describe the conditions of access to early treatment of children infected with HIV, their management on the long-term, and impact on growth, clinical and immunovirological prognosis, adherence to treatment, living conditions

DETAILED DESCRIPTION:
The CO10 EPF paediatric cohort includes therapeutic, clinical and biological detailed questionnaires. The data are collected by the doctors every three months to 2 years and then every 6 months until to 18 years or every year by a simplified questionnaire if medical follow up continues outside of a participating site.

After 18 years of age, the patients are eligibile for the ANRS CO19-Coverte cohort.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected children born to mothers included in ANRS-CO1 EPF or children under the age of 13 newly entered in care management with no prior antiretroviral therapy, whose mother was or not included in ANRS-CO1 EPF

Exclusion Criteria:

* >= 13 years
* refusal of legal representative of the child
* antiretroviral therapy started before the entry in care management
* care management for over 6 months before inclusion

Max Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Cohort of HIV-infected children born to mothers included in ANRS-CO1 EPF or children under the age of 13 newly entered in care management with no prior antiretroviral therapy, whose mother was or not included in ANRS-CO1 EPF
Sampling Method: Non-Probability Sample
Enrollment: 812 (Actual)
Dates: Start 2004-07; Primary Completion 2020-06 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Conditions of access to early treatment | At inclusion and every six months up to 18 years
  social factors (Geographical origin, living conditions, school level, age) and infection stage

SECONDARY OUTCOMES:
Puberty stage | At 8 years and every six months up to 18 years
  Tanner classification
Clinical prognosis | At inclusion and every six months up to 18 years
  Health status (lipodystrophy, metabolic abnormalities, cardiovascular diseases, encephalopathy, Developmental delay, CDC stage)
Immuno virological prognosis | At inclusion and every six months up to 18 years
  HIV RNA<50c/mL, CD4 cells count > 500 cells/mL, Genotypic resistance
Prognosis of patient coinfected by CMV or VHC | At inclusion and every six months up to 18 years
  Adverse events of treatments (complications)
Sexuality | At 15 years and every six months up to 18 years
  sexual risk behaviour (age at first intercourse, condom use at first, contraception, pregnancy, interruption of pregnancy)

CONTACTS AND LOCATIONS:
Overall Officials: Josiane WARSZAWSKI, Principal Investigator — CESP INSERM U1018
Locations (23):
- France (23):
  - CHU Angers, Angers
  - CHU Hôpital Jean Minjoz, Besançon
  - Hôpital Jean Verdier, Bondy
  - Centre Hospitalier Pellegrin, Bordeaux
  - CHU Caen, Caen
  - Hôpital Antoine Béclère, Clamart
  - Hôpital Louis Mourier, Colombes
  - Centre hospitalier Francilien Sud, Corbeil-Essonnes
  - Hôpital Bicêtre, LE Kremlin Bicëtre
  - CHR Jeanne de Flandres, Lille
  - Institut d'Hématologie et Oncologie Pédiatrique, Lyon
  - CHR Arnaud de Villeneuve, Montpellier
  - Centre Hospitalier Intercommunal, Montreuil
  - CHU Nantes Hotel Dieu, Nantes
  - CHU Hôpital de l'Archet II, Nice
  - Groupe Hospitalier Cochin Tarnier Port-Royal, Paris
  - Groupe Hospitalier Necker, Paris
  - Hôpital Robert Debré, Paris
  - Hôpital Trousseau, Paris
  - Centre Hospitalier Général- Hôpital Delafontaine, Saint-Denis
  - Hôpital Civil, Strasbourg
  - CHU Paule de Viguier, Toulouse
  - Centre Hospitalier Général, Villeneuve-Saint-Georges

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Frange P, Faye A, Avettand-Fenoel V, Bellaton E, Descamps D, Angin M, David A, Caillat-Zucman S, Peytavin G, Dollfus C, Le Chenadec J, Warszawski J, Rouzioux C, Saez-Cirion A; ANRS EPF-CO10 Pediatric Cohort and the ANRS EP47 VISCONTI study group. HIV-1 virological remission lasting more than 12 years after interruption of early antiretroviral therapy in a perinatally infected teenager enrolled in the French ANRS EPF-CO10 paediatric cohort: a case report. Lancet HIV. 2016 Jan;3(1):e49-54. doi: 10.1016/S2352-3018(15)00232-5. Epub 2015 Dec 9. PMID 26762993
- [Result] Aupiais C, Faye A, Le Chenadec J, Rouzioux C, Bouallag N, Laurent C, Blanche S, Dollfus C, Warszawski J; ANRS EPF-CO10 French Pediatric Cohort. Interruption of cART in clinical practice is associated with an increase in the long-term risk of subsequent immunosuppression in HIV-1-infected children. Pediatr Infect Dis J. 2014 Dec;33(12):1237-45. doi: 10.1097/INF.0000000000000450. PMID 24945880
- [Result] Sofeu CL, Warszawski J, Ateba Ndongo F, Penda IC, Tetang Ndiang S, Guemkam G, Makwet N, Owona F, Kfutwah A, Tchendjou P, Texier G, Tchuente M, Faye A, Tejiokem MC; ANRS-PEDIACAM Study Group. Low birth weight in perinatally HIV-exposed uninfected infants: observations in urban settings in Cameroon. PLoS One. 2014 Apr 3;9(4):e93554. doi: 10.1371/journal.pone.0093554. eCollection 2014. PMID 24705410
- [Result] Blanche S, Scott-Algara D, Le Chenadec J, Didier C, Montange T, Avettand-Fenoel V, Rouzioux C, Melard A, Viard JP, Dollfus C, Bouallag N, Warszawski J, Buseyne F. Naive T lymphocytes and recent thymic emigrants are associated with HIV-1 disease history in french adolescents and young adults infected in the perinatal period: the ANRS-EP38-IMMIP study. Clin Infect Dis. 2014 Feb;58(4):573-87. doi: 10.1093/cid/cit729. Epub 2013 Nov 18. PMID 24253249
- [Result] Avettand-Fenoel V, Blanche S, Le Chenadec J, Scott-Algara D, Dollfus C, Viard JP, Bouallag N, Benmebarek Y, Riviere Y, Warszawski J, Rouzioux C, Buseyne F. Relationships between HIV disease history and blood HIV-1 DNA load in perinatally infected adolescents and young adults: the ANRS-EP38-IMMIP study. J Infect Dis. 2012 May 15;205(10):1520-8. doi: 10.1093/infdis/jis233. Epub 2012 Mar 15. PMID 22427678
- [Result] Goetghebuer T, Le Chenadec J, Haelterman E, Galli L, Dollfus C, Thorne C, Judd A, Keiser O, Ramos JT, Levy J, Warszawski J; European Infant Collaboration Group. Short- and long-term immunological and virological outcome in HIV-infected infants according to the age at antiretroviral treatment initiation. Clin Infect Dis. 2012 Mar;54(6):878-81. doi: 10.1093/cid/cir950. Epub 2011 Dec 23. PMID 22198788
- [Result] Judd A; European Pregnancy and Paediatric HIV Cohort Collaboration (EPPICC) study group in EuroCoord. Early antiretroviral therapy in HIV-1-infected infants, 1996-2008: treatment response and duration of first-line regimens. AIDS. 2011 Nov 28;25(18):2279-87. doi: 10.1097/QAD.0b013e32834d614c. PMID 21971357
- [Result] Pursuing Later Treatment Options II (PLATO II) project team for the Collaboration of Observational HIV Epidemiological Research Europe (COHERE); Castro H, Judd A, Gibb DM, Butler K, Lodwick RK, van Sighem A, Ramos JT, Warsawski J, Thorne C, Noguera-Julian A, Obel N, Costagliola D, Tookey PA, Colin C, Kjaer J, Grarup J, Chene G, Phillips A. Risk of triple-class virological failure in children with HIV: a retrospective cohort study. Lancet. 2011 May 7;377(9777):1580-7. doi: 10.1016/S0140-6736(11)60208-0. Epub 2011 Apr 20. PMID 21511330
- [Result] Dollfus C, Le Chenadec J, Faye A, Blanche S, Briand N, Rouzioux C, Warszawski J. Long-term outcomes in adolescents perinatally infected with HIV-1 and followed up since birth in the French perinatal cohort (EPF/ANRS CO10). Clin Infect Dis. 2010 Jul 15;51(2):214-24. doi: 10.1086/653674. PMID 20536367
- [Result] Goetghebuer T, Haelterman E, Le Chenadec J, Dollfus C, Gibb D, Judd A, Green H, Galli L, Ramos JT, Giaquinto C, Warszawski J, Levy J; European Infant Collaboration group. Effect of early antiretroviral therapy on the risk of AIDS/death in HIV-infected infants. AIDS. 2009 Mar 13;23(5):597-604. doi: 10.1097/QAD.0b013e328326ca37. PMID 19194272
- [Result] Collaboration of Observational HIV Epidemiological Research Europe (COHERE) Study Group; Sabin CA, Smith CJ, d'Arminio Monforte A, Battegay M, Gabiano C, Galli L, Geelen S, Gibb D, Guiguet M, Judd A, Leport C, Dabis F, Pantazis N, Porter K, Raffi F, Thorne C, Torti C, Walker S, Warszawski J, Wintergerst U, Chene G, Lundgren J. Response to combination antiretroviral therapy: variation by age. AIDS. 2008 Jul 31;22(12):1463-73. doi: 10.1097/QAD.0b013e3282f88d02. PMID 18614870
- [Result] Warszawski J, Lechenadec J, Faye A, Dollfus C, Firtion G, Meyer L, Douard D, Monpoux F, Tricoire J, Benmebarek Y, Rouzioux C, Blanche S. Long-term nonprogression of HIV infection in children: evaluation of the ANRS prospective French Pediatric Cohort. Clin Infect Dis. 2007 Sep 15;45(6):785-94. doi: 10.1086/521165. Epub 2007 Aug 14. PMID 17712765